CLINICAL TRIAL: NCT05058378
Title: Investigation of the Correlation Between the Success of Obtaining Unilateral Spinal Anesthesia and the Measurement of Perfusion Index (pi).
Brief Title: Correlation Between Spinal Anesthesia and Perfusion Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, MEHMET DURAN, assistant professor, Adiyaman University
Other Study IDs: date:22/12/2020 ID:2020/11-20
Record Dates: First submitted 2021-09-17; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Inguinal Hernia
Keywords: spinal anesthesia, perfusion index
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: perfusion index measurement — Clip will be attached to the patient's toe for perfusion index measurement

SUMMARY:
Investigation of the correlation between the success of obtaining unilateral spinal anesthesia and the measurement of perfusion index (pi).

DETAILED DESCRIPTION:
Target sites for spinal anesthetics are spinal nerve roots and spinal cord. Differences in the anatomy of the nerve roots may explain the variability that occurs during spinal anesthesia. Spinal anesthesia is the cessation of nerve conduction for a while by injection of local anesthetic drug into the cerebrospinal fluid. It is one of the most effective and oldest regional anesthesia techniques. Unilateral spinal anesthesia, on the other hand, aims to limit the distribution of the spinal block to the operated side for all operations involving only one lower extremity. Reducing the dose of local anesthetic, pencil-point needles, injection speed, lateral decubitus position and non-isobaric anesthetic solution are the main factors in the formation of a unilateral spinal block. It requires slightly longer preparation time compared to standard spinal anesthesia, but provides fewer hemodynamic side effects with higher cardiovascular stability, increased postoperative autonomy and better patient acceptance. Perfusion index (PI) is a numerical value showing the ratio between pulsatile and nonpulsatile blood flow. PI works by measuring changes in finger peripheral perfusion via pulse oximetry. If the procedure is successful in patients undergoing spinal anesthesia, vasodilation occurs in the lower extremities due to sympathetic nerve blockage and perfusion increases. Pulse oximetry perfusion index (PI) was used in our study to indicate vasodilation associated with sympathectomy. We will examine whether the success of unilateral anesthesia in the spinal anesthesia performed in our hospital correlates with the increase of the perfusion index value measured with the finger probe, except for patient-based methods, and whether the perfusion index shows more objectively the block success than other patient-based traditional methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo lower abdominal, urogenital, lower extremity surgery
2. Patients with ASA 1-2
3. Patients aged 18-65

Exclusion Criteria:

1. Patients with ASA3-4
2. Those with peripheral vascular disease
3. Patients with a history of by-pass
4. Patients with aortic stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
perfusion index is my indicator of unilateral spinal anesthesia | 1 month
  Pulse oximetry perfusion index (PI) was used in our study to indicate vasodilation associated with sympathectomy. We will examine whether the success of unilateral anesthesia in the spinal anesthesia performed in our hospital correlates with the increase of the perfusion index value measured with the finger probe, except for patient-based methods, and whether the perfusion index shows more objectively the block success than other patient-based traditional methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to make individual participant data available to other researchers